CLINICAL TRIAL: NCT00652925
Title: Randomized, Double-Blind, Multicenter, Active Controlled Parallel Group Study to Evaluate the Efficacy and Safety of Celecoxib Suspension Compared to Naproxen Suspension in Patients With JRA
Brief Title: A Study to Evaluate the Efficacy and Safety of Celecoxib Suspension Compared to Naproxen Suspension in Patients With JRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N49-01-02-195; A3191127
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-04

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: arthritis; juvenile
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis | interventions — Celecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High Dose (Experimental)
  Interventions: Drug: Celecoxib
- Low Dose (Experimental)
  Interventions: Drug: Celecoxib
- Naproxen (Active Comparator): Control comparator, 15 mg/kg/dy target dose
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: Celecoxib — Higher dose, 6 mg/kg/dose BID
  Arms: High Dose
Drug: Celecoxib — Active drug at lower dose
  Arms: Low Dose
Drug: Naproxen — Control comparator, 15 mg/kg/dy target dose
  Arms: Naproxen

SUMMARY:
To study Celebrex versus naproxen to see if it decreases symptoms of juvenile arthritis such as pain and swelling.

ELIGIBILITY:
Inclusion Criteria:

2-18 years old with active JRA

Exclusion Criteria:

other experimental meds, recent changes in arthritis meds

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 225 (Actual)
Dates: Start 2002-10; Primary Completion 2004-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
ACR Pediatric 30 | 12 weeks

SECONDARY OUTCOMES:
Peds QOL | 12 weeks
composites of acr 30 | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (45):
- United States (24):
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Delray Beach, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Glenview, Illinois
  - Pfizer Investigational Site, Hinsdale, Illinois
  - Pfizer Investigational Site, Merrillville, Indiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Pfizer Investigational Site, Leuven, Belgium
- Brazil (2):
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Saskatoon, Saskatchewan, Canada
- Pfizer Investigational Site, Århus N, Denmark
- Pfizer Investigational Site, Vandœuvre-lès-Nancy, France
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Hanover
- Mexico (2):
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Guadalajara
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Pfizer Investigational Site, Vila Nova de Famalicão, Portugal
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Piešťany, Slovakia
- Pfizer Investigational Site, Ljubljana, Slovenia
- Spain (2):
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Valencia, Valencia
- Pfizer Investigational Site, Stockholm, Sweden

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=N49-01-02-195&StudyName=Randomized%2C%20Double-Blind%2C%20Multicenter%2C%20Active%20Controlled%20Parallel%20Group%20Study%20to%20Evaluate%20the%20Efficacy%20and%20Safety%20of%20Celecoxib%20Susp